CLINICAL TRIAL: NCT04646876
Title: Assessment Role of Mgso4 as Neuroprotective in Post Traumatic Brain Injury
Brief Title: Mgso4 as Neuroprotective in Post Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Osama Mohamed Abdelwahab (Other)
Responsible Party: Sponsor-Investigator, Osama Mohamed Abdelwahab, Professor Osama Mohamed Abdelwahab, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-142-2019
Record Dates: First submitted 2020-02-22; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Magnesium Sulphate; Traumatic Brain Injury; Brain; Injury
Keywords: Magnesium; Sulphate; double; blinded; randomized; control; study
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 2 groups, comparative
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The researcher did not know the type of medication given to the patients, placebo or treatment actually Only investigator knew the key
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention arm ( Group A ) (Active Comparator): including 30 patients Group A was given magnesium Sulphate
  Administration regimen of Mgso4 was as following:
  Initial dose: within 24 hrs of trauma 50 mg / kg / IV infusion over 1 hour. Maintenance dose: (25 mg / kg) per dose twice daily for 48 hrs.
  Interventions: Drug: Magnesium Sulfate
- Placebo arm (Group B ) (Placebo Comparator): including 30 patients Placebo control study Group B was given saline as a placebo. with the same regimen and route of administration of magnesium sulphate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — Prospective , comparative , double blind study
  Other Names: Mgso4
  Arms: intervention arm ( Group A )
Drug: Placebo — Prospective , comparative , double blind study
  Other Names: Saline
  Arms: Placebo arm (Group B )

SUMMARY:
The aim of this study is to assess the potential role of magnesium sulphate (MgSo4) as a neuroprotective agent using the Glasgow outcome scale following moderate and severe traumatic brain injury.

DETAILED DESCRIPTION:
The study is Prospective , Comparative , double-blind , placebo-controlled study with randomization

Patients with post traumatic brain injury either moderate (glasgow coma scale GCS = 9-12) or severe (GCS = 3-8) admitted in one of the neurosurgical ICU of the following centers; kasr El Aini Hospitals, Beni- Suef University Hospital or Beni- Suef General Hospital.

Study design and statistical inferences Patients with traumatic brain injury included in the study will be randomly allocated into one of two equal groups (30 patients each): -

Group (A): will receive MgSo4. Group (B): will receive normal saline as a placebo.

Each patient will receive all other standard management as indicated on individual basis (e.g. Antiepileptics, brain dehydrating measures, antibiotics, ventilatory support, or surgical intervention when deemed necessary).

The Glasgow outcome scale (GOS) will be used to categorize the outcome after 2 months as follows:

1. Death
2. Persistent vegetative state: Minimal responsiveness
3. Severe disability: Conscious but disabled; dependent on others for daily support
4. Moderate disability: Disabled but independent; can work in sheltered setting
5. Good recovery: Resumption of normal life despite minor deficits

For each patient, the following will be recorded:

1. Personal data: name, age, sex, address, tel. No.
2. Mode of trauma: fall from height, road traffic accidents, or isolated head trauma.
3. Neurological assessment on admission using the Glasgow coma score.
4. Associated injuries or neurological deficits.
5. Findings of initial CT brain, as well as follow up scans.
6. Any previous illness.

Administration :

Administration regimen of Mgso4 will be as following:

Initial dose: within 24 hrs of trauma 50 mg / kg / IV infusion over 1 hour. Maintenance dose: 25 mg / kg twice daily for 48 hrs.

In order to avoid Mgso4 toxicity, infusion of the medication (either Mgso4 or placebo) will be abruptly terminated whenever:

1. Urine output < 0.5 ml / kg / hour over 4 hours
2. Blood urea > 50 mg/ dL .
3. Fall of systolic BP < 90 mm Hg.
4. Respiratory center depression (respiratory rate less than 12 per minute).
5. Cardiac arrhythmia.
6. Loss of deep tendon reflexes.

The third supervisor will be responsible for the safety measures of the study, which will be evaluated by continuous monitoring of vital signs, arterial blood pressure (systolic, diastolic), urine output, serum chemistry.

Preparation of the drug:

The medication will be prepared by three assistants other than the researcher, one in each center where the study will be conducted.

For each patient, a set of bottles will be prepared (initial dose, and 4 maintenance doses). After preparation, each set of bottles will be labeled using the same code consisting of letters (A, B, C, D, E, F) and figures (0 to 9). Total number of codes will be 60 which is the total number of patients allocated (A0, A1, A2,....A9& B0, B1, ......B9& C1,...C9& D0-D9&E0-E9& F0-F9).

Only the second supervisor will be acquainted with the key of the code, either it is the studied treatment (Mg So4), or normal saline (placebo). He will be responsible for the random allocation of the patients, and instructing the assistants to prepare either the treatment or the placebo, and their subsequent coding. He will not be informed about the results which will be regularly followed by the first supervisor. The key will be kept hidden from the researcher who will be responsible for recording the results. The key will be disclosed only after conclusion of the study and collecting the results in order to operate the statistical analysis.

Each amp of Mgso4 (0.5 gm / 5ml) will be dissolved in 13.5 ml normal saline (at that concentration, Mgso4 will remain chemically stable for 3 months in room air). For simplicity, this will compose a unit and will be labeled as mentioned. So one unit equals 500 mg dissolved in 13.5 ml normal saline. For each patient, the number of units will be calculated according to the body weight. For example, the initial dose or the daily dose of 70 kg patient equals 7 units (70 x 50 = 3500 mg). For this patient, 3 bottles will be prepared on admission, each bottle will be labeled the same as the units, and each bottle will contain 7 units. The first bottle will be given as the initial dose, and the other two bottles will be divided to 4 equal doses, and will be given over the next 48 hrs. For placebo, the same will be done, but only using normal saline. Which is identical to Mgso4 regarding color and aspect.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with moderate (GCS = 9-12), or severe (GCS = 3-8) traumatic brain injury.

  2) Age above 12 years.

  3) Consenting for treatment within 24 hours of trauma.

Exclusion Criteria:

* 1) Non consenting patients.

  2) Persistent hypotension (BP below 90 / 60) in 1st 24 hours despite measures of resuscitation.

  3) Significant multisystem association (e.g. cord injury with spinal shock).

  4) Known case of renal failure

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Glasgow outcome scale after 2 months | 60 days from drug administration
  assessment of conscious level of the patients after 60 days of drug administration
  The Glasgow outcome scale (GOS) has been used to categorize the outcome after 2 months as follows:
  1. Death.
  2. Persistent vegetative state: Minimal responsiveness.
  3. Severe disability: Conscious but disabled; dependent on others for daily support.
  4. Moderate disability: Disabled but independent; can work in sheltered setting.
  5. Good recovery: Resumption of normal life despite minor deficits.
  Better score means that the patient conscious level is improved

CONTACTS AND LOCATIONS:
Overall Officials: Osama Awahab, professor, Principal Investigator — Faculty Of Medicine , Beni Suef University , Egypt
Locations (1):
- Faculty of medicine , Cairo university, Cairo, Egypt